CLINICAL TRIAL: NCT03406832
Title: Prevention of Coronary Slow Flow or No-Reflow During Elective Percutaneous Coronary Intervention in Patients With Acute ST-segment Elevation Myocardial Infarction
Brief Title: Prevention of Coronary Slow Flow or No-Reflow During EPCI in Patients With Acute STEMI
Acronym: NOSLOWFLOW-Ⅱ
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Collaborators: Anyang Regional Hospital (Other); Huaihe Hospital of Henan University (Other); The First Affiliated Hospital of Henan University of Science and Technology (Other); Yellow River Sanmenxia hospital (Unknown); The Peoples' Hospital of Jiaozuo City (Other); Jincheng People's Hospital (Other); The second people's Hospital of Jiyuan (Unknown); Kaifeng Central Hospital (Other); Lushan People's Hospital (Unknown); Nanyang Central Hospital (Other); The Second People's Hospital of Pingdingshan (Unknown); Shenma Medical Group General Hospital (Other); Puyang People's Hospital (Unknown); Puyang Oilfield General Hospital (Other); The First People's Hospital of Shangqiu (Unknown); Yanshi People's Hospital (Unknown); The First People's Hospital of Xinmi (Unknown); First Affiliated Hospital of Xinjiang Medical University (Other); Xinyang Central Hospital (Other); People's Hospital of Zhengzhou University (Other); Zhengzhou First People's Hospital (Unknown); Chinese Academy of Medical Sciences, Fuwai Hospital (Other); Zhengzhou Central Hospital (Other); The 99th Central Hospital of the People's Liberation Army (Unknown); Zhoukou Central Hospital (Other); The First People's Hospital of Zhumadian (Unknown); Zhumadian Central Hospital (Other)
Responsible Party: Principal Investigator, Chunguang Qiu, Director of the Department of Cardiovascular Medicine, The First Affiliated Hospital of Zhengzhou University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KS-2017-177
Record Dates: First submitted 2018-01-08; First posted 2018-01-23 (Actual); Last update posted 2019-06-07 (Actual); Status verified 2019-06

CONDITIONS: ST Segment Elevation Myocardial Infarction; Elective Percutaneous Coronary Intervention
Keywords: Prevention; Slow flow; No reflow; Nitroprusside; Tirofiban
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Nitroprusside; Tirofiban; Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nitroprusside group (Experimental): After coronary target vessel blood flow recovery by thrombus aspiration or/and balloon angioplasty (diameter ≤ 2.0mm), intracoronary infusion of Nitroprusside Sodium via guide-catheter was performed. Then repeated administration of Nitroprusside Sodium was done prior to coronary stent implantation or post dilatation.
  Interventions: Drug: Nitroprusside Sodium
- Tirofiban group (Experimental): After coronary target vessel blood flow recovery by thrombus aspiration or/and balloon angioplasty (diameter ≤ 2.0mm), intracoronary infusion of Tirofiban Hydrochloride via guide-catheter was performed.
  Interventions: Drug: Tirofiban Hydrochloride
- Control group (Placebo Comparator): After coronary target vessel blood flow recovery by thrombus aspiration or/and balloon angioplasty (diameter ≤ 2.0mm), intracoronary infusion of heparinized saline via guide-catheter was performed.
  Interventions: Drug: Heparinized saline

INTERVENTIONS:
Drug: Nitroprusside Sodium — Intracoronary infusion 50~100μg each time (repeated)
  Other Names: Experimental-1 group
  Arms: Nitroprusside group
Drug: Tirofiban Hydrochloride — Intracoronary infusion 10μg/kg for single time
  Other Names: Experimental-2 group
  Arms: Tirofiban group
Drug: Heparinized saline — Intracoronary infusion 2ml for single time
  Other Names: Control group
  Arms: Control group

SUMMARY:
Elective percutaneous coronary intervention (EPCI) is the common treatment of ST segment elevation myocardial infarction (STEMI).Slow flow / no-reflow phenomenon following EPCI in STEMI patients has been a serious and common complication that closely related to the incidence of major adverse cardiovascular events (MACE) and affected patients' prognosis. No reflow is a multi-factorial phenomenon. And its preventive and therapeutic effects are not satisfactory. This prospective randomized controlled study aimed to compare favorable effects of Nitroprusside versus Tirofiban on the prevention of slow flow / no-reflow phenomenon during EPCI.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic symptoms < 2 weeks (> 24 hours)
* Continued ischemic chest pain > 30min
* ST-segment elevation ≥ 0.1 millivolt in 2 or more contiguous leads on the 12-lead ECG or new left bundle branch block (LBBB)
* Detection of a rise of cardiac biomarker values with at least one value above the 99th percentile upper reference limit (URL)
* Elective coronary artery angiography was planned.

Exclusion Criteria:

* Emergency thrombolytic therapy was performed before elective coronary artery angiography
* Cardiogenic shock with no response to hypervolemic treatment or vasopressor
* Severe cardiomyopathy or valvular disease requiring intervention
* Coronary ectasia
* Severe heart failure
* Contraindication or allergy to antiplatelet drugs
* Contraindication or allergy to experimental drugs
* Unable to receive at least 1 year of dual antiplatelet therapy
* Active bleeding or extreme-risk for major bleeding
* Severe liver or renal failure
* Life expectancy < 1 year
* Unable or unwilling to provide informed consent
* Women of child bearing potential
* Under 18 years of age
* Hemoglobin < 90g/L
* Platelet count < 100×10^9/L
* Can not cooperate (with mental disorders or cognitive disorders)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2018-01-08 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Coronary artery flow using thrombolysis in myocardial infarction (TIMI) flow grade | 1 minute after stent implantation; 1 minute after balloon dilatation
  grade 0, no myocardial blush or contrast density; grade 1, minimal myocardial blush or contrast density; grade 2, moderate myocardial blush or contrast density but less than that obtained during angiography of a contralateral or ipsilateral noninfarct-related coronary artery; grade 3, normal myocardial blush or contrast density comparable with that obtained during angiography of a contralateral or ipsilateral noninfarct-related coronary artery.
Coronary TIMI frame count | 1 minute after stent implantation; 1 minute after balloon dilatation
  A continuous measurement assessing flow in the epicardial arteries.
Slow flow / no-reflow phenomenon | 1 minute after stent implantation; 1 minute after balloon dilatation
  Slow flow phenomenon means delayed progression or lack of contrast medium through the coronary tree.

SECONDARY OUTCOMES:
Main adverse cardiovascular and cerebrovascular events (MACCE) | at 1 day post-PCI, at follow up of 1, 3, 6,12 months post-PCI
  Death, Cardiac death, Rehospitalization (Heart failure) , Non-fatal myocardial infarction, Target vessel myocardial infarction, Target lesion revascularization, Target vessel revascularization, Ischemic-driven revascularization, Stent thrombosis, Bleeding, Cerebrovascular events, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Chunguang Qiu, Phd, Principal Investigator — The First Affiliated Hospital of Zhengzhou University
Locations (28):
- China (28):
  - Anyang District Hospital, Anyang, Henan
  - The 99th Central Hospital of the People's Liberation Army, Jiaozuo, Henan
  - The People's Hospital of Jiaozuo, Jiaozuo, Henan
  - The second people's Hospital of Jiyuan, Jiyuan, Henan
  - Huaihe Hospital of Henan University, Kaifeng, Henan
  - Kaifeng Central Hospital, Kaifeng, Henan
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Lushan People's Hospital, Lushan, Henan
  - Nanyang City Center Hospital, Nanyang, Henan
  - Pingmei Shenma Medical Group General Hospital, Pingdingshan, Henan
  - The Second People's Hospital of Pingdingshan, Pingdingshan, Henan
  - Puyang Oilfield General Hospital, Puyang, Henan
  - Puyang People's Hospital, Puyang, Henan
  - Yellow River Sanmenxia hospital, Sanmenxia, Henan
  - The First People's Hospital of Shangqiu, Shangqiu, Henan
  - The First Affiliated Hospital of Xinxiang Medical University, Xinxiang, Henan
  - Xinyang Central Hospital, Xinyang, Henan
  - Yanshi People's Hospital, Yanshi, Henan
  - Zhengzhou First People's Hospital, Zhengzhou, Henan
  - Zhengzhou Cardiovascular Hospital, Zhengzhou, Henan
  - Zhengzhou Central Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - People's Hospital of Zhengzhou, Zhengzhou, Henan
  - The First People's Hospital of Xinmi, Zhengzhou, Henan
  - Zhoukou Central Hospital, Zhoukou, Henan
  - The First People's Hospital of Zhumadian, Zhumadian, Henan
  - Zhumadian Central Hospital, Zhumadian, Henan
  - Jincheng People's Hospital, Jincheng, Shanxi

IPD SHARING:
Plan to Share IPD: No